CLINICAL TRIAL: NCT00909688
Title: Ascending Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of BLI-489 Administered Intravenously to Healthy Subjects
Brief Title: Study to Evaluate Whether BLI-489 Can be Safely Tolerated by Healthy Subjects Given Multiple Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 3219K1-1001
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — BLI-489

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): BLI-489
  Interventions: Drug: BLI-489
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: BLI-489
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
To determine the safety, tolerability, and drug absorption profile of multiple IV doses of BLI 489 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-childbearing potential (WONCBP) aged 18 to 50 years inclusive at screening;
* Body mass index (BMI) in the range of 18 to 32 kg/m2 and body weight ≥50 kg.;
* Healthy as determined by the investigator on the basis of screening evaluations;
* Calculated creatinine clearance within normal limits using the Cockcroft-Gault formula;
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history, and if a smoker must be able to abstain from smoking during the inpatient stay;
* Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study;
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease;
* Any surgical or medical condition that may interfere with the distribution, metabolism, or excretion of the investigational product;
* Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study day 1;
* History of drug abuse within 1 year before study day 1;
* Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06-05 (Actual); Primary Completion 2009-07-24 (Actual); Study Completion 2009-07-24 (Actual)

PRIMARY OUTCOMES:
Assess safety of drug given to healthy subjects by evaluating any reported adverse events (AEs), scheduled physical examinations, vital sign measurements, 12-lead ECGs, and clinical laboratory test results. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tacoma, Washington, United States